CLINICAL TRIAL: NCT00976248
Title: Phase II Study of Everolimus (RAD001) in Primary Therapy of Waldenstrom's Macroglobulinemia
Brief Title: Everolimus (RAD001) in Primary Therapy of Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Director, Bing Center, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-214
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: everolimus; RAD001; WM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): RAD001, oral, 10 mg, daily
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Taken orally once a day
  Other Names: Everolimus

SUMMARY:
The purpose of this research study is to determine the safety of RAD001(Everolimus) and the highest dose of this drug that can be given to people safely. RAD001(Everolimus) is a drug that works by preventing cells in the body from growing and dividing. Information from basic and Phase I clinical research studies suggests that RAD001 also may help to prevent tumor growth in people with relapsed or refractory lymphoma.

DETAILED DESCRIPTION:
* Participants will take RAD001 orally once a day in the morning. Each treatment cycle lasts for four weeks. Participants will receive up to 72 cycles of treatment.
* During each cycle, participants will be asked to visit the clinic for scheduled tests and exams. They will visit the clinic on the first day of each of the first three cycles, and then once every 3 cycles. During the visits, participants will have a physical exam and blood tests.. Participants may also have CT scans of the chest, abdomen and pelvis as well as a bone marrow aspirate and biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Adequate liver and renal function as outlined in the protocol
* Fasting serum cholesterol 300mg/dl or less OR 7.75mmol/L or less AND fasting triglycerides 2.5 x institutional ULN or less.
* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia as defined by consensus panel of the Second International Workshop on Waldenstrom's macroglobulinemia
* No previous therapy for WM
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of 2 times the upper limit of each institution's normal value or greater is required
* ECOG Performance status of 0-2
* Patients must have a life expectancy of at least 3 months
* Baseline platelet and absolute neutrophil as outlined in the protocol
* INR and PTT 1.5 x normalized ratio or less
* A male subject agrees to use an acceptable method for contraception for the duration of study and for 8 weeks after the last dose of the study drug
* Female subject either post-menopausal or surgically sterilized or willing to use acceptable methods of birth control for the duration of the study and for 8 weeks after the last dose of study drug

Exclusion Criteria:

* Patients experiencing symptomatic hyperviscosity and requiring plasmapheresis. This includes any patient who, in the judgement of the investigator requires urgent response and will not be eligible. These patients have hyperviscosity which includes serum IgM levels of 5000 mg/dL or greater. Symptoms may include nosebleeds, visual complications, fatigue, headaches, confusion, etc.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive any immunization with attenuated live vaccines within one week of study entry or during study period.
* Patients who have had any severe and/or uncontrolled medical conditions or other conditions that would affect their participation in the study.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001.
* Female patients that are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* Patients with known hypersensitivity to RAD001 or other rapamycins or to its excipients
* Patients with other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell of the skin
* Patients with known history of HIV seropositivity
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2016-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Treon SP, Tripsas CK, Ioakimidis L, Warren D, Patterson C, Heffner L, Eradat H, Gregory SA, Thomas S, Advani R, Baz R, Badros, Ashraf Z, Matous J, Anderson KC, Ghobrial IM Prospective, Multicenter Study of the MTOR Inhibitor Everolimus (RAD001) As Primary Therapy in Waldenstrom's Macroglobulinemia ASH Annual Meeting Abstracts 2011 118: 2951
- [Result] Treon SP, Tripsas CK, Meid K, Patterson CJ, Heffner H, Gregory SA, Thomas SK, Advani RH, Baz R, Badros AZ, Matous J, Murphy TJ, Ghobrial IM. Prospective, Multicenter Study Of The MTOR Inhibitor Everolimus (RAD001) As Primary Therapy In Waldenstrom's Macroglobulinemia Blood 2013 122:1822.
- [Derived] Treon SP, Meid K, Tripsas C, Heffner LT, Eradat H, Badros AZ, Xu L, Hunter ZR, Yang G, Patterson CJ, Gustine J, Castillo JJ, Matous J, Ghobrial IM. Prospective, Multicenter Clinical Trial of Everolimus as Primary Therapy in Waldenstrom Macroglobulinemia (WMCTG 09-214). Clin Cancer Res. 2017 May 15;23(10):2400-2404. doi: 10.1158/1078-0432.CCR-16-1918. Epub 2016 Nov 11. PMID 27836860

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: RAD001, oral, 10 mg, daily
  RAD001 : Taken orally once a day
Period: Overall Study
Arm/Group | RAD001
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of RAD001 in Patients With Previously Untreated WM
Description: Overall Response = Complete Response + Near Complete Response + Very Good Partial Response + Partial Response + Minor Response Complete Response: resolution of all symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly. A near CR (nCR) is defined as fulfilling all CR criteria in the presence of positive immunofixation test for an IgM paraprotein.
  Very Good Partial Response: > 90% reduction in serum IgM levels. Partial Response: > 50% reduction in serum IgM levels. Minor Response: 25-49% reduction in serum IgM levels Progressive Disease: greater than 25% increase in serum IgM level occurs from the lowest attained response value or progression of clinically significant disease related symptom(s).
  Stable Disease: < 25% change in serum IgM levels, in the absence of new or increasing adenopathy or splenomegaly and/or other progressive signs or symptoms of WM
Time Frame: End of Treatment, an average of 16 months
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 33
participants | 22

2. Primary Outcome: Time to Progression With Single Agent RAD001 Therapy in Previously Untreated WM.
Description: Progression is defined as a 25% increase in serum IgM from the lowest attained response value or progression of clinically significant disease related symptoms.
Time Frame: End of Treatment, an average of 16 months
Population: 13 participants were excluded from this analysis due to treatment and follow-up ending prior to progression.
Measure: Median (Full Range); unit: Months
Arm/Group | RAD001
Number analyzed (Participants) | 20
Months | 21 [1 to 64]

3. Primary Outcome: Time to Next Therapy With Single Agent RAD001 Therapy in Previously Untreated WM
Time Frame: End of follow-up, an average of 18 months
Population: 13 participants were censored due to follow-up ending prior to new therapy initiation.
Measure: Median (Full Range); unit: Months
Arm/Group | RAD001
Number analyzed (Participants) | 20
Months | 15 [1 to 69]

ADVERSE EVENTS:
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=33)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=33)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Oral ulcerations (Gastrointestinal disorders) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No